CLINICAL TRIAL: NCT00971477
Title: Evaluation of Clinical Outcomes in an Online Teledermatology Model for the Management of Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: April W. Armstrong, MD, UC Davis Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009172431
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Psoriasis
Keywords: Teledermatology; Telemedicine; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teledermatology (Experimental): Online Telemedicine Group
  Interventions: Other: Online Teledermatology Care
- Usual Care (Active Comparator): Conventional in-office care
  Interventions: Other: Conventional in Office Care

INTERVENTIONS:
Other: Online Teledermatology Care — Patients randomized to the intervention group will have their scheduled follow-up visits online via a store and forward teledermatology modality.
  Other Names: Health care service modality
  Arms: Teledermatology
Other: Conventional in Office Care — Patients randomized to the control group will have their scheduled follow-up visits via conventional in office care.
  Other Names: Health care service modality
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine if an asynchronous online model of teledermatology can achieve similar clinical outcomes as compared to conventional in-office care for the management of psoriasis. The investigators also aim to determine the effects of this online care model on patient quality of life as well as patient and physician satisfaction.

The investigators' hypotheses include the following:

1. Compared to in-person visits, the online care model will result in similar clinical improvement in psoriasis disease severity.
2. Compared to in-person visits, the online care model will result in similar improvements in quality of life.
3. Providers and subjects in the online group will achieve a similar level of overall satisfaction as those in the in-person group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent, may be men or women.
* Requiring treatment of psoriasis for medically-indicated reasons.
* Capable of giving informed consent.
* Able to have their skin imaged by themselves or by family members.

Exclusion Criteria:

* Non-English speaking individuals.
* Individuals lacking access to a digital camera and computer with internet connection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index (PASI) | Every 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: April W Armstrong, MD, Principal Investigator — UC Davis Department of Dermatology
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States